CLINICAL TRIAL: NCT00201916
Title: A Randomized Trial of a Shorter Radiation Fractionation Schedule for the Treatment of Localized Prostate Cancer
Brief Title: Shorter Radiation Schedule for the Treatment of Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: NCIC Clinical Trials Group (Network)
Responsible Party: Dr. Mark Levine, Ontario Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-1995-PR.5; CAN-OCOG-V95-0687
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate specific antigen; PSA; radiation fractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 5250 cGy in 20 fractions over 28 days
  Interventions: Procedure: 5250 cGy/20 fractions over 28 days
- 2 (Active Comparator): 6600 cGy in 33 fractions over 45 days
  Interventions: Procedure: 6600 cGy/33 fractions over 45 days

INTERVENTIONS:
Procedure: 5250 cGy/20 fractions over 28 days — see above
  Other Names: short fractionation schedule
  Arms: 1
Procedure: 6600 cGy/33 fractions over 45 days — see above
  Other Names: standard
  Arms: 2

SUMMARY:
To improve the management of patients with early stage prostate cancer.

DETAILED DESCRIPTION:
To compare the efficacy of a shorter radiation fractionation schedule to the prostate (5250 cGy/20 fractions over 28 days) with a conventional schedule (6600 cGy/33 fractions over 45 days) in men receiving radiotherapy for Stage T1a moderately or poorly differentiated, or T1b, T1c, or T2 prostate cancer. The primary outcome is local control in the prostate and secondary outcomes include toxicity, disease free survival, survival, quality of life and economics.

ELIGIBILITY:
Inclusion Criteria:

* histologic diagnosis of adenocarcinoma of the prostate with no evidence of metastatic disease to the nodes, bone or lung
* stage T1a moderately or poorly differentiated, T1b, T1c or T2 by the current UICC-TNM classification

Exclusion Criteria:

* PSA > 40 mcg/L
* previous therapy for carcinoma of the prostate other than biopsy or TURP, including patients previously on hormone therapy for treatment of their prostate cancer
* prior or active malignancy other than non-melanoma skin cancer; or colon or thyroid cancer treated a minimum of five years prior to study entry and presumed cured
* simulated volume exceeds 1000 cm3
* previous pelvic radiotherapy
* inflammatory bowel disease
* serious non-malignant disease which would preclude radiotherapy or surgical biopsy
* geographic inaccessibility for follow-up
* psychiatric or addictive disorder which would preclude obtaining informed consent or adherence to protocol
* unable to commence radiation therapy within 26 weeks of the date of last prostatic biopsy
* failure to give informed consent to participate in the study

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 936 (Actual)
Dates: Start 1995-03; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
time to PSA failure | 10 years

SECONDARY OUTCOMES:
positive biopsy at two years post radiation | see above
disease free survival | 10 years
toxicity | 10 years
quality of life | 6 years
economic | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Himu Lukka, MD, Study Chair — Juravinski Cancer Centre; Charles Hayter, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Mark Levine, MD, Principal Investigator — Ontario Clinical Oncology Group (OCOG)
Locations (16):
- Canada (16):
  - B.C. Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - B. C. Cancer Agency - Vancouver Cancer Clinic, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Dr. Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Clinic, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Toronto-Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - University Health Network -Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Lukka H, Hayter C, Julian JA, Warde P, Morris WJ, Gospodarowicz M, Levine M, Sathya J, Choo R, Prichard H, Brundage M, Kwan W. Randomized trial comparing two fractionation schedules for patients with localized prostate cancer. J Clin Oncol. 2005 Sep 1;23(25):6132-8. doi: 10.1200/JCO.2005.06.153. PMID 16135479